CLINICAL TRIAL: NCT00492869
Title: A 12-month Open-label, Randomized, Multicenter, Sequential Cohort, Dose Finding Study to Evaluate the Efficacy, Safety and Tolerability of Oral AEB071 Versus Tacrolimus in Combination With Mycophenolate Acid Sodium, Basiliximab and Corticosteroids in de Novo Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of AEB071 Versus Tacrolimus in Combination With Mycophenolate Acid Sodium, Basiliximab and Steroids in Preventing Acute Rejection After Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEB071A2207
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2016-09

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; rejection; AEB071; tacrolimus; mycophenolic; basiliximab; immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — sotrastaurin

INTERVENTIONS:
Drug: AEB071

SUMMARY:
Efficacy and safety of AEB071 in combination with mycophenolate acid sodium, basiliximab and steroids in preventing acute rejection after kidney transplantation.

ELIGIBILITY:
Inclusion:

* Male and female patients of any race 18 years or older
* Adult recipients of kidney transplant from a deceased or living donor
* Recipients of a functioning kidney within 24 hours post transplant

Exclusion:

* Need for medication prohibited by the protocol
* Patients or donors infected with Hepatitis B,C or HIV
* Patients with a history of cancer within last 5 years
* Patients with history of significant cardiac disorder
* Patients of high-risk immunological status

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Efficacy will be defined using a composite efficacy failure end point (treated biopsy proven acute rejection (BPAR), graft loss, death or loss to follow-up) between treatment and control arms

SECONDARY OUTCOMES:
Renal function assessed by calculated and measured glomerular filtration rate (GFR). Incidence of Chronic Allograft Nephropathy using biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (41):
- United States (23):
  - USC Medical Center, Los Angeles, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF, San Francisco, California
  - University of Colorado Health Science Center, Denver, Colorado
  - Lifelink, Inc., Tampa, Florida
  - U of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital Transplant Institute, Detroit, Michigan
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Comprehensive Transplant Clinic, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Dept of Internal Medicine, Cincinnati, Ohio
  - University of Toledo Health Science Campus, Toledo, Ohio
  - University of Pennsylvania Health System-Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Baylor U Medical Center, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - University of Utah, Salt Lake City, Utah
  - U of Wisconsin Hospital Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - CHU Erasme, Brussels
  - UZ Gasthuisberg, Leuven
- Canada (3):
  - Saint Joseph's Hospital, Hamilton, Ontario
  - Queen Elizabeth II, Halifax
  - Hopital Maisonneuve-Rosemont, Montreal Quebec
- Germany (6):
  - Klinikum der Humboldt Universitat Charite, Berlin
  - Universitaetsklinik Charité, Berlin
  - Staedt. Kliniken Koeln-Merheim, Cologne
  - Medizinische Hochschule Hannover, Hanover
  - Univ.-Klinikum Heidelberg, Heidelberg
  - Klinikum der Universitaet Regensburg, Regensburg
- Spain (2):
  - Hospital Juan Canalejo, A Coruña
  - Fundacion Puigvert, Barcelona
- Sweden (2):
  - Enheten f Transpl och Leverkir, SU/Sahlgrenska, Gothenburg
  - Transplantationskirurgiska mottagningen, Akademiska Sjukhuse, Uppsala
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Leicester General Hospital, Leicester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Friman S, Arns W, Nashan B, Vincenti F, Banas B, Budde K, Cibrik D, Chan L, Klempnauer J, Mulgaonkar S, Nicholson M, Wahlberg J, Wissing KM, Abrams K, Witte S, Woodle ES. Sotrastaurin, a novel small molecule inhibiting protein-kinase C: randomized phase II study in renal transplant recipients. Am J Transplant. 2011 Jul;11(7):1444-55. doi: 10.1111/j.1600-6143.2011.03538.x. Epub 2011 May 12. PMID 21564523
- See also: Results for CAEB071A2207 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2801